CLINICAL TRIAL: NCT01057212
Title: Phase II Trial of Bevacizumab and Ixabepilone for Advanced or Metastatic Non-squamous Non-small Cell Lung Cancer (NSCLC) Progressive After First-line Therapy
Brief Title: Trial of Bevacizumab and Ixabepilone for Advanced or Metastatic Non-small Cell Lung Cancer (NSCLC)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of support from pharmaceutical collaborator.
Sponsor: Providence Health & Services (Other)
Collaborators: Genentech, Inc. (Industry); Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-97B
Record Dates: First submitted 2010-01-12; First posted 2010-01-27 (Estimated); Last update posted 2015-09-07 (Estimated); Status verified 2015-09

CONDITIONS: Non-squamous Non-small Cell Lung Cancer
Keywords: advanced or metastatic non-squamous non-small cell lung cancer (NSCLC)
MeSH Terms: interventions — ixabepilone; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bevacizumab and Ixabepilone (Experimental): Bevacizumab will be administered intravenously, 10 mg/kg, every two weeks. Ixabepilone will be administered intravenously, 16 mg/m2, once weekly for 3 of 4 weeks on a 28-day schedule, to the first six patients enrolled. Ixabepilone will be administered intravenously, 20mg/m2, once weekly for 3 of 4 weeks on a 28-day schedule to the remaining 40 patients.
  Interventions: Drug: ixabepilone; Drug: bevacizumab

INTERVENTIONS:
Drug: ixabepilone — Ixabepilone will be administered intravenously, 16 mg/m2, once weekly for 3 of 4 weeks on a 28-day schedule, to the first six patients enrolled. Ixabepilone will be administered intravenously, 20mg/m2, once weekly for 3 of 4 weeks on a 28-day schedule, to the remaining 40 patients enrolled.
  Other Names: IXEMPRA®
Drug: bevacizumab — Bevacizumab will be administered intravenously, 10 mg/kg, every two weeks.
  Other Names: Avastin

SUMMARY:
This is a non-randomized, open-label, single arm phase II trial of the combination of bevacizumab and ixabepilone in patients with advanced- or metastatic non-squamous NSCLC progressive after first or second-line therapy. The main objective is to evaluate the progression-free survival in patients with advanced or metastatic non-squamous NSCLC being treated with ixabepilone and bevacizumab.

DETAILED DESCRIPTION:
The first six patients will be enrolled in a lead-in phase of the study utilizing a reduced dose of ixabepilone. Patients will be monitored for safety and toxicity. If the combination is found to be tolerable and feasible, accrual will continue with the full-dose regimen. Toxicity will be monitored in real-time by the study investigators. Should unexpected or increased toxicity be detected, trial accrual will be halted for full analysis.

Bevacizumab will be administered intravenously, 10 mg/kg, every two weeks. Ixabepilone will be administered intravenously, 16 mg/m2, once weekly for 3 of 4 weeks on a 28-day schedule, to the first six patients enrolled. Ixabepilone will be administered intravenously, 20mg/m2, once weekly for 3 of 4 weeks on a 28-day schedule, to the remaining 40 patients enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Histologic or cytologic diagnosis of advanced or metastatic non-small cell lung cancer (NSCLC), excluding squamous cell-predominant subtype. NSCLC NOS (not otherwise specified) are eligible.
* Patients must have had at least one but no more than two prior systemic chemotherapeutic regimens for metastatic disease. Prior neoadjuvant or adjuvant chemotherapy will not be included in the assessment as a prior chemotherapeutic regimen. Prior therapy with taxanes is allowed. Prior therapy with bevacizumab is allowed.
* Prior chemotherapy or therapy with investigational agents must have been completed at least 3 weeks prior to study enrollment.
* Zubrod performance status of 0 or 1.
* Patients must have measurable or evaluable disease as defined by RECIST.
* Treated brain metastases will be allowed, provided they are asymptomatic. Radiation treatment for brain metastasis must have been completed at least 2 weeks prior to enrollment. Patients must demonstrate stable symptoms and seizure control on a consistent dose of anticonvulsants for at least 2 weeks prior to enrollment. Patients must be off corticosteroids for at least 2 weeks. Treatment for brain metastases may include whole brain radiotherapy (WBRT), radiosurgery (RS; Gamma Knife, KINAC, or equivalent) or a combination as deemed appropriate by the treating physician. Patients with CNS metastases treated by neurosurgical resection or brain biopsy performed within 3 months prior to Day 1 will be excluded.
* Radiation for symptomatic lesions outside the CNS must have been completed at least 2 weeks prior to study enrollment. If measurable disease is within the radiation field, there must be evidence of clear progression (using RECIST criteria) at the time of study enrollment.
* Major surgical procedures must have been performed >28 days prior to study treatment. Portacath placement must have been performed >14 days prior to study treatment. Minor surgical procedures (fine needle aspiration, core biopsy, or mediastinoscopy) must have been performed >7 days prior to study treatment.
* Patients must have normal organ and marrow function as defined below:

  * leukocytes > 3,000/uL
  * absolute neutrophil count > 1,500/uL
  * platelets > 100,000/uL
  * total bilirubin within normal institutional limits
  * AST (SGOT)/ALT (SGPT) < 2.5 X institutional upper limit of normal
  * creatinine < 1.5 mg/dL, OR
  * calculated creatinine clearance > 40 mL/min
* Estimated life expectancy of greater than 12 weeks.
* Patients must be able to sign informed consent.
* Patients must be >18 years of age. Both men and women and members of all races and ethnic groups will be included.
* Patients must either not be of child bearing potential or, if female, have a negative serum pregnancy test within 72 hours prior to Day 1. Patients are considered not of child bearing potential if they are surgically sterile (they have undergone a vasectomy, hysterectomy, bilateral tubal ligation, bilateral oophorectomy) or they are postmenopausal with no menses for at least 12 months. Patients of childbearing potential must be willing to use adequate barrier contraception for the duration of study participation and at least 30 days after study completion.

Exclusion Criteria:

* NSCLC with predominant squamous cell histology (mixed tumors will be categorized by the predominant cell type unless small cell elements are present, in which case the patient is ineligible; sputum cytology alone is not acceptable).
* History of hemoptysis (bright red blood of 1/2 teaspoon or more per episode) within 1 month prior to Day 1.
* Known CNS disease, except for treated brain metastasis. Treated brain metastases are defined as having no evidence of progression or hemorrhage after treatment and no ongoing requirement for dexamethasone (within the last two weeks prior to Day 1), as ascertained by clinical examination and brain imaging (MRI or CT) during the screening period. Anticonvulsants (stable dose) are allowed. Treatment for brain metastases may include whole brain radiotherapy (WBRT), radiosurgery (RS; Gamma Knife, LINAC, or equivalent) or a combination as deemed appropriate by the treating physician. Patients with CNS metastases treated by neurosurgical resection or brain biopsy performed within 3 months prior to Day 1 will be excluded.
* Inability to comply with study and/or follow-up procedures.
* An investigational agent within 3 weeks of Day 1.
* Patients with greater than grade 1 neuropathy.
* Pregnant (positive pregnancy test) or lactating.
* Serious concomitant medical disorder, including active infection.
* Active second primary malignancy at the time of study enrollment.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to ixabepilone or Cremophor EL (polyoxyethylated castor oil).
* History of co-existing psychiatric illness that could impair compliance with study protocol.
* Inadequately controlled hypertension (defined as systolic blood pressure >150 and/or diastolic blood pressure > 100 mmHg on antihypertensive medications).
* Any prior history of hypertensive crisis or hypertensive encephalopathy.
* New York Heart Association (NYHA) Grade II or greater congestive heart failure.
* History of myocardial infarction or unstable angina within 6 months prior to Day 1.
* History of stroke or transient ischemic attack within 6 months prior to Day 1 of treatment.
* Significant vascular disease (e.g., aortic aneurysm, aortic dissection).
* Symptomatic peripheral vascular disease.
* Evidence of bleeding diathesis or significant coagulopathy (in the absence of therapeutic anticoagulation).
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 1 or anticipation of need for major surgical procedure during the course of the study.
* Core biopsy or other minor surgical procedure, excluding placement of a vascular access device, within 7 days prior to Day 1.
* Portacath placement within 14 days prior to Day 1.
* History of abdominal fistula or gastrointestinal perforation within 6 months prior to Day 1.
* Serious, non-healing wound, active ulcer, or untreated bone fracture.
* Proteinuria at screening as demonstrated by either:

  * Urine protein: creatinine (UPC) ratio ≥ 1.0 at screening OR
  * Urine dipstick for proteinuria ≥ 2+ (patients discovered to have ≥2+ proteinuria on dipstick urinalysis at screening should undergo a 24 hour urine collection and must demonstrate ≤ 500 mg of protein in 24 hours to be eligible).
* Known hypersensitivity to any component of bevacizumab.
* Prior discontinuation of bevacizumab due to treatment-related toxicity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2010-02; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
progression-free survival | at week 8, week 16, and every 8 weeks until disease progression or removal from study

SECONDARY OUTCOMES:
To evaluate the overall response rate using RECIST criteria | at week 8, week 16, and every 8 weeks until disease progression or removal from study
toxicities associated with treatment combination in advanced non-squamous NSCLC | all treatment days and every 2 months post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Sanborn, MD, Principal Investigator — Providence Health & Services
Locations (1):
- Providence Portland Medical Center, Portland, Oregon, United States